CLINICAL TRIAL: NCT01936012
Title: Bioequivalence Study of 10 mg Lisinopril Tablets (Lisinopril 10 mg) Produced by PT Dexa Medica in Comparison With The Innovator Tablets (Zestril® 10 mg, PT Boehringer Ingelheim Indonesia, Indonesia, Under License From Astra Zeneca UK Ltd.)
Brief Title: Bioequivalence Study of Two Formulations of 10 mg Lisinopril Tablet Under Fasting Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BE.258/EQL/2012
Record Dates: First submitted 2013-09-01; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Lisinopril; Bioequivalence; Bioavailability; Pharmacokinetic; Angiotensin-converting enzyme inhibitor
MeSH Terms: interventions — Lisinopril

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisinopril 10 mg tablets of PT Dexa Medica (Experimental): Each tablet contains 10.89 mg lisinopril dihydrate that equal to 10 mg lisinopril. A single dose of lisinopril tablet of PT Dexa Medica was given to each of study subjects.
  Interventions: Drug: Lisinopril 10 mg tablets of PT Dexa Medica
- Lisinopril 10 mg tablets of PT Boehringer Ingelheim Indonesia (Active Comparator): Each tablet contains 10.89 mg lisinopril dihydrate that equal to 10 mg lisinopril. A single dose of lisinopril tablet of PT Boehringer Ingelheim Indonesia was given to each of study subjects.
  Interventions: Drug: Lisinopril 10 mg tablets of PT Boehringer Ingelheim Indonesia

INTERVENTIONS:
Drug: Lisinopril 10 mg tablets of PT Dexa Medica — Each tablet contains 10.89 mg of lisinopril dihydrate that equal to 10 mg lisinopril. Test product was given as a single dose, under the procedure as described in the Section: Detailed description of the study.
  Other Names: Test Product: Lisinopril 10 mg tablets of PT Dexa Medica
  Arms: Lisinopril 10 mg tablets of PT Dexa Medica
Drug: Lisinopril 10 mg tablets of PT Boehringer Ingelheim Indonesia — Each tablet contains 10.89 mg of lisinopril dihydrate that equal to 10 mg lisinopril. Reference product was given as a single dose, under the procedure as described in the Section: Detailed description of the study.
  Other Names: Reference product: Zestril® 10 mg, produced by PT Boehringer Ingelheim Indonesia, under license from Astra Zeneca UK Ltd..
  Arms: Lisinopril 10 mg tablets of PT Boehringer Ingelheim Indonesia

SUMMARY:
The present study was conducted to find out whether the bioavailability of 10 mg lisinopril tablets produced by PT Dexa Medica was equivalent to the tablets produced by the innovator (Zestril® 10 mg, PT Boehringer Ingelheim Indonesia, Indonesia, under license from Astra Zeneca UK Ltd.)

DETAILED DESCRIPTION:
This was a randomized, single-blind, two-period, two-sequence, cross-over study under fasting condition. The participating subjects were required to have an overnight fast and in the next morning were given orally one tablet of the test drug (Lisinopril 10 mg, produced by PT Dexa Medica) or one tablet of the reference drug (Zestril® 10 mg, PT Boehringer Ingelheim Indonesia, Indonesia, under license from Astra Zeneca UK Ltd.).

Blood samples were drawn immediately before taking the drug (control), and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 36, and 48 hours after drug administration. Seven days after the first drug administration (washout period), the procedure was repeated using the alternate drug.

The pharmacokinetic parameters, including AUCt, AUCinf, Cmax, t max, and t1/2, were determined from plasma concentrations of lisinopril, using liquid chromatography with tandem mass spectrometry detection (LC-MS/MS) method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects.
* Aged 18 - 55 years inclusive.
* Non-smokers or moderate smokers (less than 10 cigarettes per day).
* Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study.
* Body mass index within 18 to 25 kg/m2.
* Vital signs (after 10 minutes rest) were within the following ranges:

  * systolic blood pressure 110 - 120 mmHg
  * diastolic blood pressure 70 - 80 mmHg
  * pulse rate 60 - 90 bpm

Exclusion Criteria:

* Personal/family history of allergy or hypersensitivity or contraindication to lisinopril or allied drugs.
* Pregnant or lactating women.
* Any major illness or clinically significant ongoing chronic medical illness in the past 90 days.
* Any clinically significant abnormality of liver function test (ALT, AP, total bilirubin >= 1.5 ULN).
* Any clinically significant abnormality of renal function test (serum creatinine concentration > 1.4 mg/dL).
* Positive hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV.
* Clinically significant hematology abnormalities.
* Clinically significant electrocardiogram (ECG) abnormalities.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study drug.
* Past history of anaphylaxis or angioedema.
* History of drug or alcohol abuse within 12 months prior to screening.
* Participation in any clinical trial within the past 90 days.
* History of any bleeding or coagulative disorders.
* History of difficulty with donating blood or accessibility of veins in left or right arm.
* A donation or loss of 500 mL (or more) of blood within 3 months before the study's first dosing day.
* Intake of any prescription or non-prescription drugs, food supplements, or herbal medicines within 14 days of the study's first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the last observed quantifiable concentration (AUCt) of lisinopril | 48 hours
  Relative bioavailability (primarily measured by AUCt and AUCinf) between two lisinopril 10 mg tablet formulations (test and reference formulations) was assessed under fasting condition. AUCt was determined from plasma concentration of lisinopril.
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) of lisinopril | 48 hours
  Relative bioavailability (primarily measured by AUCt and AUCinf) between two lisinopril 10 mg tablet formulations (test and reference formulations) was assessed under fasting condition. AUCinf was determined from plasma concentration of lisinopril.

SECONDARY OUTCOMES:
The peak plasma concentration (Cmax) of lisinopril | 48 hours
  Relative bioavailability (secondarily measured by Cmax) between two lisinopril 10 mg tablet formulations (test and reference formulations) was assessed under fasting condition. Cmax was determined from plasma concentration of lisinopril.
Time needed to achieve the peak plasma concentration (t max) of lisinopril | 48 hours
  Relative bioavailability (secondarily measured by t max) between two lisinopril 10 mg tablet formulations (test and reference formulations) was assessed under fasting condition. t max was determined from plasma concentration of lisinopril.
The elimination half-life (t1/2) of lisinopril | 48 hours
  Relative bioavailability (secondarily measured by t1/2) between two lisinopril 10 mg tablet formulations (test and reference formulations) was assessed under fasting condition. t1/2 was determined from plasma concentration of lisinopril.

CONTACTS AND LOCATIONS:
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia